CLINICAL TRIAL: NCT06459076
Title: Application of Transnasal Humidified Rapid-insufflation Ventilatory Exchange (THRIVE) in Burn Children With Suspected Difficult Airway：A Single-center, Randomized Controlled Study
Brief Title: Application of THRIVE in Burn Children With Suspected Difficult Airway
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shuxiu Wang (Other)
Responsible Party: Sponsor-Investigator, Shuxiu Wang, Principal Investigator, The First Affiliated Hospital of Air Force Medicial University
Organization: The First Affiliated Hospital of Air Force Medicial University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1stAHAirforceMedicalU
Record Dates: First submitted 2024-06-01; First posted 2024-06-14 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Intubation; Difficult or Failed
Keywords: THRIVE; burn children; airway; intubation
MeSH Terms: interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Routine Care group (No Intervention): After induction of general intravenous anesthesia, 100% oxygen mask ventilation was used for pre-oxygenation, wait 2-3 min to vecuronium take effect and reaching end-expiratory oxygen saturation > 90%, the Optiflow THRIVETM system nasal plug is placed in the proper position, but without oxygen supply, and the tracheal intubation is started.
- THRIVE group (Experimental): After induction of general intravenous anesthesia, 100% oxygen mask ventilation was used for pre-oxygenation, wait 2-3 min to vecuronium take effect and reaching end-expiratory oxygen saturation > 90%, Immediately after ceasing assisted ventilation, the age-appropriate nasal prongs were applied and weight-specific high flow rates delivered using the(Transnasal humidified rapid-insufflation ventilatory exchange, THRIVE) Optiflow THRIVE TM system. The flow rates applied were as follows: 0-15 kg, 2 litres kg-1 min-1；15-30 kg, 35 litres min-1; 30-50 kg, 40 litres min-1; and>50 kg, 50 litres min-1,and the tracheal intubation is started
  Interventions: Device: Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE)

INTERVENTIONS:
Device: Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) — Immediately after ceasing assisted ventilation, before intubation the age-appropriate nasal prongs were applied and weight-specific high flow rates delivered using the Optiflow THRIVETM system. The flow rates applied were as follows: 0-15 kg, 2 litres kg-1 min-1；15-30 kg, 35 litres min-1; 30-50 kg, 40 litres min-1; and>50 kg, 50 litres min-1.
  Arms: THRIVE group

SUMMARY:
In order to improve intubation conditions in burn children, our aim is to investigate the efficacy of transnasal humidified rapid-insufflation ventilatory exchange technique（THRIVE) in children aged between 0 and 18 years who with head, face, and neck injuries by fire, scalding, chemical, electric,explosions, and others. We hypothesise that THRIVE increases first attempt success without hypoxemia in intubation of children and compared with routine practice.

Does the THRIVE can prolong apnoea time and delay the onset of desaturation to increase the success rate of the first tracheal intubation without desaturation?

Researchers will compare THRIVE group with Routine care group to see successful intubation on the first attempt without desaturation.

Participants will received intravenous anesthesia induction, followed by 2-3 minutes preoxygenation, before intubation, the mask was removed from the children's face and a THRIVE nasal plug was placed. During intubation, the Routine care group had no oxygen supply,and the THRIVE group will be maintained throughout the apnoeic period with selected flow rates during intubation attempts.

DETAILED DESCRIPTION:
The incidence of burns is four times higher in children than in adults: burn injuries account for about 25% of all paediatric hospitalisations. Approximately 70 percent of children who attend hospital with burns or scalds are less than five years of age. The most common cause is hot liquids. Direct heat and steam injury to the upper airway can lead to marked swelling of the face, tongue, epiglottis, and glottic opening, resulting in airway obstruction,especially for these who burned with head,face and neck. Dressings and nasogastric tubes may make face mask seal difficult, facial wounds may be painful, and exudate and topical antibiotics may make for a slippery surface and difficult for anesthesiologist to holding the mask during preoxygenation phase. However,In children, awake intubation is not a viable option. Therefore, intubation is often attempted after Rapid Sequence Intubation (RSI) by set up a vein line after inhalation anesthesia in the operating room. But the lower functional residual capacity and greater metabolic demand of children made the onset of desaturation in apnoeic children occurs much faster than in adults at induction of anaesthesia and is known to be age dependent. If the desaturation occurs, oxygen mask is often required to manually assist ventilation, until SPO2 recovery after another attempt to intubation. Attempting more than two tracheal intubations in children with difficult endotracheal intubation is associated with a high failure rate and increased incidence of complications.

Preoxygenation does not supply an ongoing gas exchange and therefore there is an urgent need for newer methods to continue improved oxygenation during the apnoeic phase.Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) has potential in pre-oxygenation for RSI anaesthesia since it provides high-flow humidified oxygen through nasal cannulae and allows continued peri-laryngoscopy oxygen delivery during apnoea.

Therefore, investigator propose the hypothesis that children with head, face, and neck burns or thermal scalds use THRIVE during endotracheal intubation after anesthesia induction, It can prolong the safe apnoea oxygenation time and increase the success rate of the first intubation without SPO2 decrease ≤90%.

No sedative was applied before patients entering the operating room. All patients were put in the"sniffing" position with a 2-2.5 cm pad placed under shoulder in order to maintain upper airway patency. Intravenous anesthesia was induced with fentanyl 2ug/kg-1 and propofol 2-3mg/kg-1 and vecuronium 0.1 mg/kg-1, respectively,(for children without or with difficulty in set up vein line, 8% sevoflurane was inhaled, and after I.V. access was established,Sevoflurane were discontinued,followed by Intravenous induction), (The preoxygenation phase is defined as the period in preparation for intubation where oxygen is delivered to The patient to maximize oxygen concentration in the functional residual capacity of The lung), and wait 2-3 min for vecuronium to takes effect after reaching end-expiratory oxygen saturation > 90%,the manual ventilation is stopped and according to different groups, different intervention was performed. Routine care group: after stopping manual ventilation, the inestigators immediately removed the mask and placed the nasal plug in place but without oxygen supply, and the anesthesiologist began to intubation; THRIVE group: after stopping manual ventilation, the investigators immediately ceasing assisted ventilation, the age-appropriate nasal prongs were applied and weight-specific high flow rates delivered using The Optiflow THRIVETM system. The flow rates applied were as follows: 0-15kg, 2litres KG-1 Min-1; 15-30kg, 35litres Min-1; 30-50kg, 40litres Min-1; and & GT; 50kg, 50litres Min-1,and start to tracheal intubation.

If SPO2 ≤ 90% appears during intubation, then perform manual ventilation immediately until SPO2 returned to 100% endotracheal intubation was performed again and recorded as second attempt intubation.

Monitoring of anesthetic depth was not possible because The surgical site involved The head and face.

ELIGIBILITY:
Inclusion Criteria:

* < 18 years
* ASA Grade I ~ III
* Children with head, face and neck scald or burn or flame or electrical c hemical or other

Exclusion Criteria:

* Refusal or failure to sign an informed consent
* Proposed to transnasal intubation
* Fracture of the nasal bone, nasal bleeding, nasal deformity or obstruction
* Tracheotomy status or severe head, face and neck burn or burn scar (difficult airway)
* Unsuitable for rapid sequence induction
* Basicranial fracture
* Cyanotic congenital heart defect
* At risk of malignant hyperthermia
* And is participating in other clinical studies

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of successful intubation on the first attempt without physiological instability | through study completion, an average of 2 years
  Physiological instability is defined as SPO2≤90% at any time after induction of anesthesia until endotracheal intubation is completed.
  A successful first attempt intubation is defined as a successful intubation at first attempt without any desaturation (SpO2≤90% or saturation difference ≥10% for who after pre-oxygenation SpO2 cannot reach 100%).
  Successful intubation was defined as completion of the intubation attempt with correct placement of the endotracheal tube, as confirmed by the detection of expired carbon dioxide with a colorimetric detector.

SECONDARY OUTCOMES:
Rate of hypoxemia; time to and duration of desaturation during the intubation attempt; the duration and number of intubation attempts; nadir SPO2 and heart rate during intubation attempt. | through study completion, an average of 2 years
  Time to desaturation was defined as the time in seconds from ceasing assisted ventilation until the SpO2 first dropped below 90%.
  The duration of desaturation the time from the initial drop below 90% until the SpO2 rose above 100% again.
  An intubation attempt was defined as the insertion of the laryngoscope blade beyond the patient's lips until its removal from the patient's mouth, whether or not an attempt was made to insert an endotracheal tube. or where there is a change in operator during the procedure even if the device is not removed.
  Intubation time was defined as the time from the start of laryngoscopy, when the blade was introduced between the teeth, until the first breath with the tracheal tube in place, verified by capnography.

CONTACTS AND LOCATIONS:
Overall Officials: shuxiu wang, PH.D, Principal Investigator — The Xijing Hospital of Air Force Military Medical University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Legrand M, Barraud D, Constant I, Devauchelle P, Donat N, Fontaine M, Goffinet L, Hoffmann C, Jeanne M, Jonqueres J, Leclerc T, Lefort H, Louvet N, Losser MR, Lucas C, Pantet O, Roquilly A, Rousseau AF, Soussi S, Wiramus S, Gayat E, Blet A. Management of severe thermal burns in the acute phase in adults and children. Anaesth Crit Care Pain Med. 2020 Apr;39(2):253-267. doi: 10.1016/j.accpm.2020.03.006. Epub 2020 Mar 5. PMID 32147581
- [Result] Jeschke MG, Herndon DN. Burns in children: standard and new treatments. Lancet. 2014 Mar 29;383(9923):1168-78. doi: 10.1016/S0140-6736(13)61093-4. Epub 2013 Sep 11. PMID 24034453
- [Result] Bittner EA, Shank E, Woodson L, Martyn JA. Acute and perioperative care of the burn-injured patient. Anesthesiology. 2015 Feb;122(2):448-64. doi: 10.1097/ALN.0000000000000559. PMID 25485468
- [Result] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Result] Patel A, Nouraei SA. Transnasal Humidified Rapid-Insufflation Ventilatory Exchange (THRIVE): a physiological method of increasing apnoea time in patients with difficult airways. Anaesthesia. 2015 Mar;70(3):323-9. doi: 10.1111/anae.12923. Epub 2014 Nov 10. PMID 25388828
- [Result] Humphreys S, Lee-Archer P, Reyne G, Long D, Williams T, Schibler A. Transnasal humidified rapid-insufflation ventilatory exchange (THRIVE) in children: a randomized controlled trial. Br J Anaesth. 2017 Feb;118(2):232-238. doi: 10.1093/bja/aew401. PMID 28100527
- [Result] Hodgson KA, Owen LS, Kamlin COF, Roberts CT, Newman SE, Francis KL, Donath SM, Davis PG, Manley BJ. Nasal High-Flow Therapy during Neonatal Endotracheal Intubation. N Engl J Med. 2022 Apr 28;386(17):1627-1637. doi: 10.1056/NEJMoa2116735. PMID 35476651
- [Result] Overmann KM, Boyd SD, Zhang Y, Kerrey BT. Apneic oxygenation to prevent oxyhemoglobin desaturation during rapid sequence intubation in a pediatric emergency department. Am J Emerg Med. 2019 Aug;37(8):1416-1421. doi: 10.1016/j.ajem.2018.10.030. Epub 2018 Oct 18. PMID 30401594
- [Result] Kerrey BT, Rinderknecht AS, Geis GL, Nigrovic LE, Mittiga MR. Rapid sequence intubation for pediatric emergency patients: higher frequency of failed attempts and adverse effects found by video review. Ann Emerg Med. 2012 Sep;60(3):251-9. doi: 10.1016/j.annemergmed.2012.02.013. Epub 2012 Mar 15. PMID 22424653
- See also: PubMed ID:32147581 — https://pubmed.ncbi.nlm.nih.gov/32147581/
- See also: PubMed ID:24034453 — https://pubmed.ncbi.nlm.nih.gov/24034453/
- See also: PubMed ID:25485468 — https://pubmed.ncbi.nlm.nih.gov/25485468/
- See also: PubMed ID:26705976 — https://pubmed.ncbi.nlm.nih.gov/26705976/
- See also: PubMed ID:25388828 — https://pubmed.ncbi.nlm.nih.gov/25388828/
- See also: PubMed ID:28100527 — https://pubmed.ncbi.nlm.nih.gov/28100527/
- See also: PubMed ID:35476651 — https://pubmed.ncbi.nlm.nih.gov/35476651/
- See also: PubMed ID:30401594 — https://pubmed.ncbi.nlm.nih.gov/30401594/
- See also: PubMed ID:22424653 — https://pubmed.ncbi.nlm.nih.gov/22424653/